CLINICAL TRIAL: NCT00295126
Title: Use of Autologous Platelet Concentrate in Pre-Implantation Reconstruction of Maxilla.
Brief Title: REPI : a Randomized Open Label Trial Evaluating the Use of APC in Pre-Implantation Reconstruction of Maxilla
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Etablissement Français du Sang (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 01 12
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Jaw, Edentulous; Tooth Loss; Maxillary Diseases
Keywords: Edentulous; Tooth Loss; APC; Autologous platelet concentrate
MeSH Terms: conditions — Jaw, Edentulous; Tooth Loss; Maxillary Diseases; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cellular therapy : Autologous platelet concentrate (APC)

SUMMARY:
This is a randomized open label trial that evaluates the efficacy of an autologous platelet concentrate (APC) in pre-implantation reconstruction of maxilla.

The sinus occlusion will be performed under general anaesthetic. On one side by the usual technique with hipbone transplant, the other side will be restored with APC mixed with autologous bone tissue removed from the surgery site.

The side selection will be determined by the randomization.

DETAILED DESCRIPTION:
Rational

Maxillary Edentulous is one of the more frequent handicaps that cause many problems for dental prosthesis. Dental implants are currently the most convenient solution but require sufficient bone sinus height.

The filling of the sinus can be made by two ways :

* Either with autologous bone removed from hipbone or cranial bone. This method has several drawbacks such as the multiplicity of the surgery sites.
* Or with alloplasty materials that are subject to uncertain osseointegration and that are very expensive.

The aim of this study is to show the interest of an autologous platelet concentrate (APC) in this surgery. We will use the osteogenic property of platelets associated with a small quantity of spongy bone removed from the surgery site.

It has been previously demonstrated that platelets contain growth factors, in particular PDGF (platelet derivated growth factors), TGF-α1 and 2 (transforming growth factors) and IGF-1 (insulin like growth factor). These molecules have receptors on spongy bone, enhance mitosis, osteoblast differentiation, angiogenesis and induce the inhibition of osteoclats.

Method :

The sinus filling will be performed under general anaesthetic. On one side by the usual technique with hipbone transplant, the other side will be restored with APC mixed with autologous bone tissue removed from the surgery site.

The side selection will be determined by the randomization. For each patient a waiting period of 6 months is required before dental implants.

Twenty patients will be enrolled in this single-centre study with a follow-up of one year.

Main objective :

- To demonstrate that the osteogenesis with APC mixed with a small quantity (1 to 2 cm2) of autologous bone tissue removed from the surgery site, has a sufficient quality to allow the dental implants.

Secondary Objectives :

* To compare the osteogenesis with the current procedure (hipbone transplant)
* To estimate the kinetic of osteogenesis using successive radiography.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* ASA1 class of anesthetic risk
* SA3 or SA4 of the Misch classification

Exclusion Criteria:

* Smoker
* Progressive sinusal lesion or previous history of maxillary sinusitis
* Previous history of maxillary surgery
* Hemopathy
* Contraindication to cytapheresis
* Progressive cardiopathy
* Severe cerebellar arteriopathy
* Infectious state
* Thrombopenia < 150 g/l controlled by citrate
* Serology : antibody anti-HVC, anti-HIV 1 & 2, anti HTLV 1 & 2 positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-05; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Radiological outcome measure : the bone height under the sinus on the two sides.

SECONDARY OUTCOMES:
Radiological outcome measure : the bone density
Clinical outcome measure : assessment of the alveolar crest quality, possible orals complications, and complications at the removal site.
Histological outcome measures : with bone core boring at the implant site.
All these measurements will be matched for each patient on both sides.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Bettega, Dr, Principal Investigator — Univesity Grenoble Hospital, Stomatology Department
Locations (1):
- University Hospital of Grenoble, Grenoble, Isere, France

REFERENCES:
- [Background] Robiony M, Polini F, Costa F, Politi M. Osteogenesis distraction and platelet-rich plasma for bone restoration of the severely atrophic mandible: preliminary results. J Oral Maxillofac Surg. 2002 Jun;60(6):630-5. doi: 10.1053/joms.2002.33107. PMID 12022097
- [Background] Carlson ER. Bone grafting the jaws in the 21st century: the use of platelet-rich plasma and bone morphogenetic protein. Alpha Omegan. 2000 Aug-Sep;93(3):26-30. PMID 11212572
- [Background] Kassolis JD, Rosen PS, Reynolds MA. Alveolar ridge and sinus augmentation utilizing platelet-rich plasma in combination with freeze-dried bone allograft: case series. J Periodontol. 2000 Oct;71(10):1654-61. doi: 10.1902/jop.2000.71.10.1654. PMID 11063400
- [Background] Lebeau J, Savariaux C, Perrier P, Bettega G, Raphael B. [Functional evaluation of intraoral reconstructive surgery. A valuable tool: articulatory evaluation of the acoustic signal]. Rev Stomatol Chir Maxillofac. 2000 Apr;101(2):60-4. French. PMID 10859754